CLINICAL TRIAL: NCT06349577
Title: Optimizing Pulsatility During Cardiopulmonary Bypass to Reduce Acute Kidney Injury: Randomized Controlled Trial
Brief Title: Optimizing Pulsatility During Cardiopulmonary Bypass to Reduce Acute Kidney Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-0921; 5K23HL151882 (NIH)
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Hemolysis; Thrombocytopenia; Surgery
MeSH Terms: conditions — Acute Kidney Injury; Hemolysis; Thrombocytopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-pulsatile blood flow (Active Comparator): Non-pulsatile blood flow during cardiopulmonary bypass
  Interventions: Other: Non-pulsatile blood flow
- Pulsatile blood flow (Active Comparator): Pulsatile blood flow during cardiopulmonary bypass
  Interventions: Other: Pulsatile blood flow

INTERVENTIONS:
Other: Non-pulsatile blood flow — Non-pulsatile blood flow generated by constant centrifugal pump flow rate during cardiopulmonary bypass
  Arms: Non-pulsatile blood flow
Other: Pulsatile blood flow — Pulsatile blood flow generated by variable centrifugal pump flow rate during cardiopulmonary bypass
  Arms: Pulsatile blood flow

SUMMARY:
The objective is to determine the effectiveness of pulsatile flow during cardiopulmonary bypass to reduce the incidence of acute kidney injury after cardiac surgery. Investigators will also evaluate the safety and impact of pulsatile flow on clinical outcomes compared to non-pulsatile flow during cardiopulmonary bypass.

DETAILED DESCRIPTION:
Non-pulsatile and pulsatile blood flow during cardiopulmonary bypass for cardiac surgery are both considered standard of care and allow surgeons to operate on the heart without movement. Pulsatile cardiopulmonary bypass produces variations in blood flow to produce a pulse similar to a normal beating heart. Non-pulsatile and pulsatile blood flow during cardiopulmonary bypass are approved as safe and effective ways to provide perfusion during cardiac surgery, but it is unknown whether there are differences in clinical outcomes after surgery. Acute kidney injury is common after cardiac surgery and may be caused by inadequate perfusion during cardiopulmonary bypass.

Specific Aim: The purpose of this study is to determine the effectiveness of pulsatile blood flow during cardiopulmonary bypass to reduce the incidence of acute kidney injury after cardiac surgery compared to non-pulsatile blood flow.

Hypothesis: Pulsatile blood flow during cardiopulmonary bypass will reduce the incidence of acute kidney injury after cardiac surgery compared to non-pulsatile blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Scheduled for elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria

* Emergency procedures
* Scheduled for heart or lung transplantation
* Scheduled for ventricular assist device implantation
* Use of the Medtronic Elongated Once-Piece Arterial Cannula
* Diagnosed with sepsis
* Diagnosed with delirium
* Experiencing hemodynamic instability (heart rate > 100 and systolic blood pressure < 90)
* Requiring mechanical circulatory support
* Requiring vasoactive medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | From intensive care unit admission after surgery up to 7 days
  Stage 1 (mild), 2 (moderate), or 3 (severe) acute kidney injury according to the Kidney Disease Improving Global Outcomes creatinine criteria (stage 1 = 1.5 to 1.9 times baseline or greater than or equal to 0.3 milligrams per deciliter increase in serum creatinine, stage 2 = 2.0 to 2.9 times baseline in serum creatinine, stage 3 = 3.0 times baseline or increase in serum creatinine greater than or equal to 4.0 milligrams per deciliter or initiation of renal replacement therapy

SECONDARY OUTCOMES:
Acute kidney injury risk score | On admission to the intensive care unit after surgery up to 24 hours after intensive care unit arrival
  Demirjian Perioperative Laboratory Test-Based Prediction Model for Moderate to Severe Acute Kidney Injury After Cardiac Surgery in percent predicted risk
Red blood cell units transfused | After cardiopulmonary bypass up to 24 hours after intensive care unit arrival
  Number of allogenic red blood cell units transfused after cardiopulmonary bypass
Platelet nadir | On admission to the intensive care unit after surgery up to 7 days
  Lowest platelet count after cardiopulmonary bypass
Discontinuation rate of cardiopulmonary bypass mode | During cardiopulmonary bypass
  Discontinuation rate of pulsatile or non-pulsatile cardiopulmonary bypass mode
30-day mortality | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  All cause mortality

OTHER OUTCOMES:
Myocardial infarction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Myocardial infarction by clinical diagnosis
Stroke | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Stroke by clinical diagnosis
Renal failure requiring renal replacement therapy | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New diagnosis of renal failure requiring renal replacement therapy
Re-exploration for bleeding | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Surgical re-exploration for bleeding
Sepsis | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Diagnosed by positive blood culture
New onset atrial fibrillation | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Clinical diagnosis of new onset atrial fibrillation
Duration of mechanical ventilation | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Duration of mechanical ventilation
Post-operative delirium | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative determined by the Confusion Assessment Method for the Intensive Care Unit
Post-operative hospital length of stay | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative hospital length of stay
New requirement for mechanical circulatory support | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New requirement for mechanical circulatory support
Intra-operative red blood cell transfusion in units | During the intra-operative time period, up to 12 hours
  Intra-operative red blood cell transfusion in units
Post-operative red blood cell transfusion in units | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative red blood cell transfusion in units
Post-operative platelet transfusion in units | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative platelet transfusion in units
Post-operative plasma transfusion in units | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative plasma transfusion in units
Post-operative cryoprecipitate transfusion in units | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Post-operative cryoprecipitate transfusion in units
Intra-operative platelet transfusion in units | During the intra-operative time period, up to 12 hours
  Intra-operative platelet transfusion in units
Intra-operative plasma transfusion in units | During the intra-operative time period, up to 12 hours
  Intra-operative plasma transfusion in units
Intra-operative cryoprecipitate transfusion in units | During the intra-operative time period, up to 12 hours
  Intra-operative cryoprecipitate transfusion in units
New onset of acute lung injury | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  Diagnosis of acute lung injury by PaO2 to FiO2 ratio ≤ 300
New onset of left ventricular systolic dysfunction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New onset of left ventricular systolic dysfunction determined by a LV ejection fraction <50%
New onset of right ventricular systolic dysfunction | From intensive care unit admission after surgery to hospital discharge, up to 30 days
  New onset of right ventricular systolic dysfunction determined by a tricuspid annular plane systolic excursion less than 16 mm

CONTACTS AND LOCATIONS:
Overall Officials: Nathan J Clendenen, MD, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demirjian S, Bashour CA, Shaw A, Schold JD, Simon J, Anthony D, Soltesz E, Gadegbeku CA. Predictive Accuracy of a Perioperative Laboratory Test-Based Prediction Model for Moderate to Severe Acute Kidney Injury After Cardiac Surgery. JAMA. 2022 Mar 8;327(10):956-964. doi: 10.1001/jama.2022.1751. PMID 35258532
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Tan A, Newey C, Falter F. Pulsatile Perfusion during Cardiopulmonary Bypass: A Literature Review. J Extra Corpor Technol. 2022 Mar;54(1):50-60. doi: 10.1182/ject-50-60. PMID 36380831